CLINICAL TRIAL: NCT01609608
Title: Whole-Body Vibration for Functional Constipation: A Single-Center, Single-Blinded, Randomized, Controlled Trial
Brief Title: Whole-Body Vibration for Functional Constipation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Changhua Christian Hospital (Other)
Responsible Party: Principal Investigator, Tsung Ju Wu, Medical doctor, Changhua Christian Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 091004
Record Dates: First submitted 2012-05-28; First posted 2012-06-01 (Estimated); Last update posted 2012-06-01 (Estimated); Status verified 2012-05

CONDITIONS: Constipation
MeSH Terms: conditions — Constipation

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- vibration (Experimental)
  Interventions: Procedure: whole body vibration
- placebo (Placebo Comparator)
  Interventions: Procedure: whole body vibration

INTERVENTIONS:
Procedure: whole body vibration — to deliver mechanical oscillation to individuals at various frequencies, amplitudes, and accelerations for different durations. This technique has been applied for years to enhance strength, and improve bone mineral density and balance

SUMMARY:
1. Aim: The aim of this trial was to determine whether whole-body vibration (WBV) induced via a non-invasive oscillation platform could improve symptoms and health-related quality of life (HRQOL) in patients with chronic functional constipation.
2. Methods: A single-blinded, randomized, control trial was performed in a single Hospital in Taiwan. Patients diagnosed with chronic functional constipation, as per the Rome III diagnostic criteria were included and randomized to either the WBV treatment or no treatment (control) group. The treatment group received six 15-minute sessions of WBV therapy over a two-week period. Patients received vibrations of 2 mm in amplitude at a frequency of 12 Hz. The primary outcome was assessed by the constipation severity instrument (CSI). The secondary outcome was improvements in HRQOL.

ELIGIBILITY:
Inclusion Criteria:

* met the Rome III criteria of constipation

Exclusion Criteria:

* pregnant
* cardiovascular disease
* cerebrovascular disease
* recently undergone major surgery
* hypothyroidism
* depressive disorder.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2009-10; Primary Completion 2010-10 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
change from baseline in constipation severity instrument (CSI) at 2 weeks | baseline (day 1), the completion of the trial (day 14)

SECONDARY OUTCOMES:
change from baseline in health-related quality of life (HRQOL) at 2 weeks | baseline (day 1), the completion of the trial (day 14)

CONTACTS AND LOCATIONS:
Locations (1):
- Changhua Christian hospital, Changhua, Taiwan, Taiwan

REFERENCES:
- [Result] Prisby RD, Lafage-Proust MH, Malaval L, Belli A, Vico L. Effects of whole body vibration on the skeleton and other organ systems in man and animal models: what we know and what we need to know. Ageing Res Rev. 2008 Dec;7(4):319-29. doi: 10.1016/j.arr.2008.07.004. Epub 2008 Aug 12. PMID 18762281
- [Derived] Wu TJ, Wei TS, Chou YH, Yang CP, Wu CL, Chen YC, Liu SY. Whole-body vibration for functional constipation: a single-centre, single-blinded, randomized controlled trial. Colorectal Dis. 2012 Nov;14(11):e779-85. doi: 10.1111/codi.12021. PMID 22966839